CLINICAL TRIAL: NCT07084714
Title: Impact of Moderate Aerobic Exercise on Menstrual Cycle Symptoms in Sedentary Women
Brief Title: Moderate Aerobic Exercise for Managing Menstrual Cycle Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Colorado Springs (Other)
Responsible Party: Principal Investigator, Marissa Baranauskas, Assistant Professor, University of Colorado, Colorado Springs
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOVE
Record Dates: First submitted 2025-07-09; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Premenstrual Syndrome; Menstrual Cycle; Menstrual Distress (Dysmenorrhea); Menstrual Bleeding, Heavy
Keywords: menstrual cycle; premenstrual syndrome; dysmenorrhea
MeSH Terms: conditions — Premenstrual Syndrome; Dysmenorrhea; Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-hormonal contraceptive users (Experimental): Women who report regular menstrual periods every 21-35 days and have not used hormonal or non-hormonal (i.e., intrauterine device) contraceptives in the past 6 months.
  Interventions: Behavioral: Moderate Aerobic Exercise
- Hormonal contraceptive users (Experimental): Women who are taking a combined oral contraceptive (i.e., those that contain a form of progesterone and estrogen) for at least the past 6 months.
  Interventions: Behavioral: Moderate Aerobic Exercise

INTERVENTIONS:
Behavioral: Moderate Aerobic Exercise — Participants will complete moderate intensity aerobic exercise for 30 minutes per session, progressing from three to five days per week to meet the minimum recommended aerobic physical activity guideline of 150 minutes per week set by the American College of Sports Medicine (ACSM) over two menstrual cycles. Moderate intensity is defined as maintaining a heart rate within 40-59% heart rate reserve and a rate of perceived exertion of 11-14 "light to somewhat hard" on the Borg 6-20 scale.

SUMMARY:
The goal of this clinical trial is to evaluate the impact of moderate aerobic exercise on menstrual symptom management in sedentary women both using and not using hormonal contraceptives. The main questions it aims to answer are:

Is there a reduction in physical and/or psychological menstrual cycle related symptom burden with participation in moderate aerobic exercise for sedentary women using and not using hormonal contraceptives?

Is there a difference in physical and/or psychological menstrual cycle related symptom burden between hormonal contraceptive and non-hormonal contraceptive users?

Is a moderate aerobic exercise intervention more effective in reducing physical and/or psychological menstrual related symptom burden for sedentary women using or not using hormonal contraceptives?

Participants will:

* Have their body composition assessed using dual energy X-ray absorptiometry pre and post exercise intervention.
* Complete a Menstrual Symptom Index (MSi) to report daily menstrual cycle related symptom burden in addition to the Premenstrual Symptom Screening Tool (PSST) and Heavy Menstrual Bleeding (HMB) questionnaire monthly.
* Utilize an at-home monitor to test urinary luteinizing hormone, estrone-3-glucuronide, and pregnanediol glucuronide approximately 10 times per month and report menstrual cycle length.
* Record physical activity habits by continuously wearing a wrist-based accelerometer and chest-strap heart rate monitor during planned aerobic exercise sessions and complete the International Physical Activity Questionnaire (IPAQ) monthly.
* Maintain their usual sedentary activity habits for one menstrual cycle followed by completion of an exercise intervention designed to progress individuals to meet minimum recommended aerobic physical activity guidelines of 150 minutes per week set by the American College of Sports Medicine for two menstrual cycles.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal (defined as having regular menstrual periods every 21-35 days)
* either not using hormonal or non-hormonal contraceptives (i.e., intrauterine device) for the past 6 months OR using combined oral contraceptives (i.e., those that contain progesterone and estrogen) for at least the past 6 months
* not currently pregnant or trying to become pregnant
* sedentary lifestyle (score of "low activity/inactive" assessed using the IPAQ)
* have self reported menstrual cycle symptoms (symptoms reported on the PSST or MSi)
* do not have a medical diagnosis or signs/symptoms of diabetes, cardiovascular, or renal disease and are able to participate in moderate intensity physical activity without physician clearance

Exclusion Criteria:

* becoming physically active defined as scoring higher than "low activity/inactive" on the IPAQ during the first month of the study
* non compliance with instructions provided for the moderate aerobic exercise intervention (i.e., not adhering to predetermined intensity heart rate targets) or miss more than 25% of exercise sessions in either intervention month
* becoming pregnant during enrollment
* being diagnosed with a cardiovascular, metabolic, or renal disease that would require physical clearance to participate in moderate intensity aerobic physical activity
* begin using hormonal or non-hormonal (i.e., intrauterine devices) contraceptives if assigned to the arm not using hormonal contraceptives
* either begin a different type of contraceptive or discontinue combined hormonal contraceptive use if assigned to the hormonal contraceptive arm

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Menstrual Symptom Index (MSi) scores | Baseline, 1 month, and 2 months
  The MSi asks participants to report the intensity they are experiencing 18 menstrual related symptoms on a scale ranging from 0 = "do not feel at all" to 3 = "intense." A score of 0 indicates no symptom burden and 54 the maximum symptom burden.
Change from baseline in Premenstrual Symptoms Screening Tool (PSST) - Symptoms | Baseline, 1 month, 2 month
  The PSST has participants report the intensity which they experience 14 premenstrual symptoms on a scale ranging from 0 = "not at all" to 3 = "intense". A score of 0 reflects no premenstrual symptom burden and a score of 42 indicates maximal premenstrual symptom burden.
Change from baseline in Premenstrual Symptoms Screening Tool (PSST) - Quality of Life | Baseline, 1 month, 2 months
  The PSST asks participants to report the severity by which premenstrual symptoms affect 4 functional aspects of life related to work, relationships with coworkers and family, and home responsibilities on a scale ranging from 0 = "not at all" to 3 = "severe". A score of 0 indicates no interference and 12 maximal interference.

OTHER OUTCOMES:
Urinary luteinizing hormone (LH) | Baseline, month 1, month 2
  mIU/mL
Urinary pregnanediol glucuronide (PdG) | Baseline, 1 month, 2 months
  ug/mL
Urinary estrone-3-glucuronide (E3G) | Baseline, month 1, month 2
  ng/mL

CONTACTS AND LOCATIONS:
Locations (1):
- William J. Hybl Sports Medicine and Performance Center, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No